CLINICAL TRIAL: NCT02653209
Title: TriMaster: Randomised Double-Blind Crossover Study of a DPP4 Inhibitor, SGLT2 Inhibitor and Thiazolidinedione as Third Line Therapy in Patients With Type 2 Diabetes Who Have Suboptimal Glycaemic Control on Dual Therapy With Metformin and a Sulphonylurea
Brief Title: TriMaster: Study of a DPP4 Inhibitor, SGLT2 Inhibitor and Thiazolidinedione as Third Line Therapy in Patients With Type 2 Diabetes.
Acronym: TriMaster
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other); NHS Tayside (Other Government); University of Dundee (Other); University of Glasgow (Other); Newcastle University (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1603221; 2015-002790-38 (EudraCT Number); 12039221 (Registry Identifier: ISRCTN); MR/N00633X/1 (Other Grant/Funding Number: Medical Research Council, UK)
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Stratification; Biomarkers; Pharmacogenetics; SGLT2 inhibitors; Thiazolidinediones; DPP4 inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Canagliflozin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin - DPP4i (Experimental)
  Interventions: Drug: Sitagliptin - DPP4i
- Canagliflozin - SGLT2i (Experimental)
  Interventions: Drug: Canagliflozin - SGLT2i
- Pioglitazone - TZD (Experimental)
  Interventions: Drug: Pioglitazone - TZD

INTERVENTIONS:
Drug: Sitagliptin - DPP4i — DPP4 inhibitor 100mg supplied as over-encapsulated hard capsule shell to be taken orally, once a day for 16 weeks in addition to existing prescribed oral diabetes therapy.
  Other Names: Januvia
  Arms: Sitagliptin - DPP4i
Drug: Canagliflozin - SGLT2i — SGLT2 inhibitor 100mg supplied as over-encapsulated hard capsule shell to be taken orally, once a day for 16 weeks in addition to existing prescribed oral diabetes therapy.
  Other Names: Invokana
  Arms: Canagliflozin - SGLT2i
Drug: Pioglitazone - TZD — Thiazolidinedione 30mg supplied as over-encapsulated hard capsule shell to be taken orally, once a day for 16 weeks in addition to existing prescribed oral diabetes therapy.
  Other Names: Actos
  Arms: Pioglitazone - TZD

SUMMARY:
The aim of this project is to identify subgroups of patients with type 2 diabetes that respond well or poorly to particular drugs based on particular clinical characteristics such as their weight or kidney function, to enable better targeting of treatment for a particular individual.

This study will test 2 hypotheses of drug response supported by routine clinical and trial data. 600 patients with type 2 diabetes who have suboptimal glycaemic control on dual oral therapy will be recruited to a randomised double-blind crossover study of a DPP4 inhibitor, SGLT2 inhibitor and thiazolidinedione. Each patient will take each study drug in addition to their existing treatment for four months at a time. At the end of each treatment the patient's glucose control will be measured and information about their experience of the drug will be collected.

DETAILED DESCRIPTION:
The study is a phase 4 randomised double-blind crossover study of a DPP4 inhibitor, SGLT2 inhibitor and thiazolidinedione as third line therapy in patients with Type 2 diabetes who have suboptimal glycaemic control on dual therapy with metformin and a sulphonylurea.

600 patients aged 30-80 who have been on stable doses of 2 classes of therapy (not including the trial IMPs or GLP1-agonist) for at least 3 months with HbA1c >58mmol/mol (7.5%) will receive three double-blinded third-line non-injectable therapies. On recruitment into the study participants will have underlying pathophysiology assessed in a mixed-meal tolerance test (MMTT) and samples will be collected for baseline analysis and storage for future biomarker analysis and discovery. Participants will then receive 16 weeks of each over-encapsulated blinded therapy in random order.

At the end of each treatment period, fasting blood will be taken to measure glycaemic response (HbA1c), fasting glucose and insulin concentrations trough drug levels and to confirm continued eligibility. Weight, blood pressure and. data about patient experience will also be collected including perceived side effects, preparedness to remain on therapy, psychological health and health related quality of life.

At the end of the study, patient treatment preference will be recorded after feeding back to the patient for each of the 3 therapies their HbA1c, weight change, frequency of hypoglycaemias, any patient reported side effects and the patient's verdict on each therapy will be recorded. Each participant will be asked which treatments they would take long term and the reason for their preference.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes
* Age ≥30 and ≤80
* Currently treated with two classes of oral glucose-lowering therapy (given either as separate or combined medications), that do not include a DPP4-inhibitor, a SGLT2-inhibitor or a thiazolidinedione.
* Diabetes duration ≥12months
* No change in diabetes treatment (new treatments or dose change) within previous 3 months
* HbA1c > 58mmol/mol (7.5%) and ≤110mmol/mol (12.2%) - confirmed at screening visit
* eGFR ≥ 60mls/min/1.73m² - confirmed at screening visit
* Able and willing to give informed consent

Exclusion Criteria:

* Changes in glucose-lowering therapy or dose within last 3 months
* HbA1c ≤ 58mmol/mol (7.5%) or >110mmol/mol (12.2%)
* eGFR <60mls/min/1.73m².
* Diabetes duration <12 months
* ALT >2.5 x upper limit of the assay normal range or known liver disease, specifically >30 μmol/L that is associated with other evidence of liver failure.
* Insulin treated within the last 12 months
* Limb ischaemia shown by absence of both pulses in one or both feet.
* Currently treated with corticosteroids
* Currently treated with rifampicin, gemfibrozil, phenytoin and carbamazepine
* Active infection (any infection requiring antibiotics at present)
* Foot ulcer requiring antibiotics within previous three months
* Recent (within 3 months) significant surgery or planned surgery (excluding minor procedures)
* Acute cardiovascular episode (angina, myocardial infarction, stroke, transient ischemic episode) occurring within the previous 3 months
* History of heart failure
* Current use of loop diuretic therapy (Furosemide or Bumetanide)
* History of bladder carcinoma
* Current/ongoing investigation for macroscopic haematuria
* History of Diabetic Ketoacidosis
* History of pancreatitis
* Pregnant, breastfeeding or planning a pregnancy over the study period
* Concurrent Participation on another Clinical Trial of an Investigational Medicinal Product, where the IMP is currently being taken, or without sufficient washout period* and without consultation with the CTIMP research team.
* Unable or unwilling to give informed consent

  * Sufficient washout period = five times the half-life of the IMP / potential IMP if involving a placebo / longest half-life if a trial includes more than one drug

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
On treatment HbA1c in obese patients (BMI >30kgm-2), compared to non-obese patients | 16 weeks
  Outcome measure will test hypothesis that patients with insulin resistance, characterised clinically by a raised BMI (>30 kg/m2), compared to non-obese patients, will:
  1. Respond well to pioglitazone, a thiazolidinedione that works as an insulin sensitiser.
  2. Respond less well to sitagliptin, a DPP4i, which works through stimulating endogenous insulin secretion post-prandially.
On treatment HbA1c in patients with an eGFR <90 mls/min/1.73m2 compared to patients with an eGFR >90 mls/min/1.73m2. | 16 weeks
  Outcome measure will test hypothesis that patients with modestly reduced estimated glomerular filtration rate (eGFR 60-90 mls/min/1.73m2), compared to those with eGFR >90 mls/min/1.73m2, will:
  1. Respond poorly to canagliflozin, a SGLT2 inhibitor, which works through inhibiting the active reabsorption of glucose in the proximal tubule, as the reduced eGFR will reduce the glucose-lowering efficacy.
  2. Respond well to sitagliptin, a DPP4i that is renally cleared, as the reduced eGFR will increase plasma DPP4i concentrations.

SECONDARY OUTCOMES:
Patient preference | 48-54 weeks (3 x 16 weeks of therapy)
  Patient treatment preference of study drug within hypothesised strata and overall
Prevalence of side effects | 48-54 weeks (3 x 16 weeks of therapy)
  Prevalence of side effects within hypothesised strata and for specific drugs, to include: weight gain, hypoglycaemia, oedema, genital tract infection and discontinuation of therapy
HbA1c on therapy against predefined test of gender heterogeneity | 16 weeks
  Predefined test of gender heterogeneity with pilot data suggesting females are likely to show an improved response relative to males for pioglitazone.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hattersley, Principal Investigator — University of Exeter / Royal Devon & Exeter NHS Trust
Locations (1):
- Exeter Clinical Research Facility, Exeter, United Kingdom

REFERENCES:
- [Derived] Shields BM, Angwin CD, Shepherd MH, Britten N, Jones AG, Sattar N, Holman R, Pearson ER, Hattersley AT. Patient preference for second- and third-line therapies in type 2 diabetes: a prespecified secondary endpoint of the TriMaster study. Nat Med. 2023 Feb;29(2):384-391. doi: 10.1038/s41591-022-02121-6. Epub 2022 Dec 7. PMID 36477734
- [Derived] Shields BM, Dennis JM, Angwin CD, Warren F, Henley WE, Farmer AJ, Sattar N, Holman RR, Jones AG, Pearson ER, Hattersley AT; TriMaster Study group. Patient stratification for determining optimal second-line and third-line therapy for type 2 diabetes: the TriMaster study. Nat Med. 2023 Feb;29(2):376-383. doi: 10.1038/s41591-022-02120-7. Epub 2022 Dec 7. PMID 36477733
- [Derived] Angwin C, Jenkinson C, Jones A, Jennison C, Henley W, Farmer A, Sattar N, Holman RR, Pearson E, Shields B, Hattersley A; MASTERMIND consortium. TriMaster: randomised double-blind crossover study of a DPP4 inhibitor, SGLT2 inhibitor and thiazolidinedione as second-line or third-line therapy in patients with type 2 diabetes who have suboptimal glycaemic control on metformin treatment with or without a sulfonylurea-a MASTERMIND study protocol. BMJ Open. 2020 Dec 21;10(12):e042784. doi: 10.1136/bmjopen-2020-042784. PMID 33371044

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT02653209/SAP_000.pdf